CLINICAL TRIAL: NCT04211870
Title: Effects of Photobiomodulation in Children With Down Syndrome and Possible Sleep Bruxism: Protocol For A Randomized, Controlled, Blind, Clinical Trial
Brief Title: Effects of Photobiomodulation in Children With Down Syndrome and Possible Sleep Bruxism
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DownSyndrome
Record Dates: First submitted 2019-12-19; First posted 2019-12-26 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Sleep Bruxism
MeSH Terms: conditions — Sleep Bruxism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Intervention (Experimental): Treatment with LED clusters.
  Interventions: Radiation: LED clusters

INTERVENTIONS:
Radiation: LED clusters — Each LED board contains six (6) LEDs with a wavelength of 660nm and a duration of seven (7) minutes in each muscle. The treatment was carried out in a total of four (4) sessions, one (1) session per week.

SUMMARY:
The main characteristic of an individual with Trisomy 21 (T21), commonly known as Down Syndrome (DS), is muscular hypotonia, a characteristic that mainly affects the masticatory and oropharyngeal muscles, resulting in impairments in speech, swallowing, breathing and chewing, in addition to pain, noise and/or degeneration in the temporomandibular joints (TMJ), therefore, developing bruxism. The gold standard for the treatment and control of bruxism is the rigid plate, however, there is difficulty in developing treatment in children and adolescents with T21, therefore, photobiomodulation is a non-invasive intervention alternative already consolidated as an excellent option for modulation in muscle tissues. This study sought to evaluate the efficacy and safety of non-invasive intervention with red LED clusters for the control of bruxism in children and adolescents diagnosed with Down Syndrome. The present study is characterized as a pilot study, composed of individuals of both sexes, aged 4 to 17 years old, attended at the UNINOVE integrated health clinic and diagnosed with Down syndrome and bruxism. The treatment was carried out in a total of four sessions, one session per week, where in each session the LED plates were applied and post-application electromyographic collection was carried out.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with a diagnosis of Down syndrome
* Four to 17 years of age
* Bruxism, based on parental reports of the occurrence of grinding the teeth, incisal and/or occlusal tooth wear following the criteria of the American Academy of Sleep Medicine (AASM) and the questionnaire for the evaluation of bruxism validated by Serra Negra et al. (2014) and a systematic review performed by Manfredini et al. (2013).

Exclusion Criteria:

* Use of muscle relaxant
* Temporomandibular disorder
* Undergoing other therapy for bruxism
* Other associated neurological diseases
* Cognitive deficit that impedes understanding the evaluations.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of electromyography of masticatory muscles | Baseline and immediately after each the procedure.
  The activation of the masseter muscles (right and left) and anterior temporalis (right and left) has analyses of electrical activities that were collected by means of the BTS TMJOINT electromyograph from BTS Engineering with 6 channels, 4 of which are used, containing a bioelectric signal amplifier, wireless data transmission (wireless system) and disposable bipolar surface electrodes (Ag/AgCl - Medical Trace®) with 10 mm in diameter. The EMG signal was amplified with a gain of 2000 times and filtered within a frequency of 20-450 Hz. The impedance and common rejection mode of the equipment are >1015 Ω//0.2 pF and 60/10Hz 92 dB.

SECONDARY OUTCOMES:
Orofacial Evaluation Through NOT-S (score from 0 to 12) | Baseline and immediately after each the procedure.
  The following functions are addressed during the interview: (I) sensory function, (II) breathing, (III) habits, (IV) chewing and swallowing, (V) drooling and (VI) dryness of the mouth. The following functions are evaluated during the physical examination: (1) face at rest, (2) nose breathing, (3) facial expression, (4) masticatory muscle and jaw function, (5) oral motor function and (6) speech. For the evaluation of orofacial dysfunction during the clinical examination, the participants will be asked to perform tasks for each item in accordance with the illustrated manual. Each item has criteria for the respective function. A "YES" response or task the meets the criteria for compromised function will be scored 1 point, indicating dysfunction in the respective domain. A "NO" response or task that does not meet the criteria will be scored zero. The total is the sum of the points of all domains and ranges from 0 to 12, with higher scores denoting greater orofacial disfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Nove de Julho University, São Paulo, Brazil

REFERENCES:
- [Derived] Salgueiro MDCC, Silva T, Motta LJ, Horliana ACRT, Goncalves MLL, Gomes AO, Pinto MM, Bortoletto CC, Altavista OM, Deana AM, Silva DFTD, Santos EM, Castelo PM, Fernandes KPS, Mesquita-Ferrari RA, Bussadori SK. Effects of Photobiomodulation in Children with Down Syndrome and Possible Sleep Bruxism: Protocol For A Randomized, Controlled, Blind, Clinical Trial: Study protocol clinical trial (SPIRIT compliant). Medicine (Baltimore). 2020 Apr;99(17):e19904. doi: 10.1097/MD.0000000000019904. PMID 32332670